CLINICAL TRIAL: NCT03707457
Title: Phase I Protocol to Assess Safety of Biomarker-Driven Therapy Using Selective Immune Activators in Combination With Anti-PD-1 (Nivolumab) in Patients With First Recurrence of Glioblastoma
Brief Title: Biomarker-Driven Therapy Using Immune Activators With Nivolumab in Patients With First Recurrence of Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding/material support withdrawn
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J17154; IRB00129944 (Other: JHM IRB)
Record Dates: First submitted 2018-10-10; First posted 2018-10-16 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Nivolumab; spartalizumab; MK-4166; epacadostat; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Nivolumab + anti-GITR (Experimental): Patients receive nivolumab intravenously (IV) over 30 minutes and anti-GITR intravenously (IV) over 30 minutes on Day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nivolumab; Drug: Anti-GITR Monoclonal Antibody MK-4166
- Arm B: Nivolumab + IDO1 inhibitor (Experimental): Patients receive nivolumab intravenously (IV) over 30 minutes on Day 1 and IDO1 inhibitor daily by mouth. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nivolumab; Drug: IDO1 inhibitor INCB024360
- Arm C: Nivolumab + Ipilimumab (Experimental): Patients receive nivolumab intravenously (IV) over 30 minutes and ipilimumab intravenously (IV) over 90 minutes on Day 1. Courses repeat every 21 days for up to 4 doses. After ipilimumab is discontinued, courses of nivolumab repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Patients receive nivolumab intravenously (IV) over 30 minutes on Day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Other Names: anti-PD1
Drug: Anti-GITR Monoclonal Antibody MK-4166 — Patients receive anti-GITR intravenously (IV) over 30 minutes on Day 1 of the first cycle of nivolumab after arm assignment. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Other Names: anti-GITR
  Arms: Arm A: Nivolumab + anti-GITR
Drug: IDO1 inhibitor INCB024360 — Patients receive IDO1 inhibitor by mouth daily beginning on Day 1 of the first cycle of nivolumab after arm assignment. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Arms: Arm B: Nivolumab + IDO1 inhibitor
Drug: Ipilimumab — Patients receive ipilimumab intravenously (IV) over 90 minutes on Day 1 of the first cycle of nivolumab after arm assignment. Courses repeat every 21 days for up to 4 doses in the absence of disease progression or unacceptable toxicity.
  Arms: Arm C: Nivolumab + Ipilimumab

SUMMARY:
This research is being done to test if it is safe to give nivolumab with targeted immunotherapy drugs for recurrent glioblastoma (GBM), a type of brain tumor. The study doctors believe that giving immunotherapy drugs that match the biomarkers in a tumor will help the immune system fight the tumor. Tumor tissue collected during surgery will be tested for certain biomarkers to determine which immunotherapy might best target the tumor.

The combination immunotherapy arms include:

Arm A: Nivolumab + anti-GITR Arm B: Nivolumab + IDO1 inhibitor Arm C: Nivolumab + Ipilimumab

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

1. To determine safety of each of the following study agents, anti-GITR, IDO1 inhibitor, and ipilimumab, in combination with nivolumab (BMS-936558) flat dose in patients with first recurrence of GBM.

SECONDARY OBJECTIVES

1. To estimate toxicity
2. To estimate progression-free survival
3. To estimate overall survival
4. To evaluate pain for patients undergoing the treatment of anti-GITR, IDO1 inhibitor, and ipilimumab, in combination with nivolumab.

EXPLORATORY OBJECTIVES

1. To characterize the immune response during and after treatment as measured by immunohistochemistry, and other T cells etc. in peripheral blood
2. To characterize the pharmacodynamic and genomic activity in tumor tissue as target inhibition
3. To characterize radiographic response
4. Genetic characterization of correlative samples

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically proven glioblastoma or gliosarcoma which is progressive or recurrent following radiation therapy with or without temozolomide.
* Patient must be in first recurrence of glioblastoma following radiation therapy with or without temozolomide. Patients with previously grade 3 astrocytoma who after first recurrence after radiotherapy with or without temozolomide are found to have GBM are eligible. Patients with previously grade 3 glioma found to have conclusively progressed to GBM at the time screening tissue is taken are eligible. Patients who have received Gliadel wafers during their initial surgery are eligible.
* Patient must be undergoing repeat surgery that is clinically indicated as determined by their care providers, where a significant debulking or a gross total surgical resection of the contrast-enhancing area is intended.
* Patient must consent to our acquiring tumor tissue removed before, during, or after the study, if it becomes available.
* Patient must be able to undergo MRI of the brain with gadolinium.
* Patient must have recovered from severe toxicity of prior therapy. An interval of at least 12 weeks must have elapsed since the completion of radiation therapy or placement of Gliadel wafers, and at least 6 weeks must have elapsed from the last dose of temozolomide (TMZ) before starting Nivolumab. Patients must stop using the Optune device prior to starting nivolumab. No prior therapies are allowed other than radiation, temozolomide, Optune device, and Gliadel wafers (placed during the first surgery at diagnosis of high grade glioma (HGG)).
* Patients must be 18 years of age or older.
* Patients must have a Karnofsky Performance Status (KPS) ≥ 60% (i.e. the patient must be able to care for himself/herself with occasional help from others).
* Patients must have the following organ and marrow function:
* Absolute lymphocyte count ≥ 500/mcl
* Absolute neutrophil count ≥ 1,500/mcl
* Platelets ≥ 100,000/mcl
* Hemoglobin ≥ 9 g/dl
* Total bilirubin ≤ institutional upper limit of normal (except for patients with Gilberts' syndrome who must have normal direct bilirubin)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional upper limit of normal
* Creatinine ≤ institutional upper limit of normal OR Creatinine clearance ≥ 60 ml/min/1.73m2 for patients with creatinine levels above institutional normal
* activated partial thromboplastin time (APTT) or partial thromboplastin time (PTT) ≤ 1.5 x institutional upper limit of normal
* Patient must be able to provide written informed consent.
* Women of childbearing potential (WOCBP) must agree to have a negative serum pregnancy test within -7 days prior to treatment start. Women of childbearing potential must agree to use non-hormonal (due to induction of Cyp3a4) (barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment, and through at least 5 months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Males who are sexually active with WOCBP must agree to use a condom during penile vaginal intercourse for the duration of treatment with study treatment plus 7 months after the last dose of the study treatment (i.e., 90 days [duration of sperm turnover] plus the time required for nivolumab to undergo approximately 5 half-lives). This criteria applies to azoospermic males as well.
* Patient must not have another malignancy unless disease free for ≥ 5 years. Curatively treated basal or squamous cell carcinoma of the skin, totally excised melanoma of stage IIA or lower, low- or intermediate-grade localized prostate cancer (Gleason sum ≤7), and curatively-treated carcinoma in situ of the cervix, breast, or bladder are allowed regardless.

Exclusion Criteria:

* Patient is/has received any other investigational agent(s).
* Patient has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to IO agents used in this study.
* Patient has active or a known history of known or suspected autoimmune disease. (Subjects with Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, and skin disorders (vitiligo, psoriasis, or alopecia) not requiring systemic treatment, are permitted to enroll.
* Patient has a condition requiring systemic treatment with either corticosteroids (other than for brain tumor management, cerebral edema or hypothalamic-pituitary dysfunction) or other immunosuppressive medications within 14 days of study entry.
* Patient has evidence of significant mass effect.
* Patient has evidence of significant hematologic, renal, or hepatic dysfunction. (NOTE: Patients with underlying hepatocellular disease should be given careful risk/benefit consideration prior to enrollment).
* Patient has a known history of any chronic hepatitis as evidenced by the following:

  * Positive test for hepatitis B surface antigen (HBsAg)
  * Positive test for qualitative hepatitis C viral load (by PCR) (Note: Subjects with positive hepatitis C antibody and negative quantitative hepatitis C by PCR are eligible. History of resolved hepatitis A virus infection is not an exclusion criterion.)
  * History of alcoholic or non-alcoholic steatohepatitis (NASH), auto-immune hepatitis, or previous grade 3-4 drug-related hepatitis, or any form of chronic liver disease.
* Patient has a confirmed history of encephalitis or meningitis in the year prior to signing informed consent.
* Patients with uncontrolled or significant cardiovascular disease including, but not limited to, any of the following are ineligible:

  * Myocardial infarction or stroke/transient ischemic attack (TIA) within the 6 months prior to consent
  * Uncontrolled angina within the 3 months prior to consent
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
  * QTc prolongation > 480 msec
  * History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, myocarditis, congestive heart failure with New York Heart Association (NYHA) functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, deep venous thrombosis, etc.)
  * Cardiovascular disease-related requirement for daily supplemental oxygen
* Patient has another uncontrolled intercurrent illness including, but not limited to, ongoing or active infection that requires systemic antibacterial, antiviral or antifungal therapy < 7 days prior to the first dose of study drug, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible.
* Patient is pregnant or breastfeeding.
* Patient has a known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Participants with a personal or family (i.e., in a first-degree relative) history of cytochrome b5 reductase deficiency (previously called methemoglobin reductase deficiency) or other diseases that put them at risk of methemoglobinemia. All participants will be screened for methemoglobin levels prior to arm assignment.
* Patient has a history of G6PD deficiency or other congenital or autoimmune hemolytic disorders
* Patient has/had prior organ or tissue allograft.
* Patient has a history of life-threatening toxicity related to prior immune therapy.
* Patient has quantitative or qualitative G6PD assay results suggesting underlying G6PD deficiency.
* Patient has blood methemoglobin > ULN, assessed in an arterial or venous blood sample or by cooximetry.
* Patient has a history or presence of hypersensitivity or idiosyncratic reaction to methylene blue.
* Patient has a history of serotonin syndrome.
* Participants with active interstitial lung disease (ILD) or pneumonitis or with recent history of ILD or pneumonitis requiring steroids (excluding radiation pneumonitis)
* Patient has active interstitial lung disease (ILD) or pneumonitis or with recent history of ILD or pneumonitis requiring steroids (excluding radiation pneumonitis).
* Patient has condition(s) known to interfere significantly with the absorption of oral medication, as per investigator judgement.
* Patient is taking any prohibited medications unless discontinued at least 10 days prior to initiation of therapy (unless otherwise specified in the protocol).
* Patient is taking any restricted medications that per investigator judgement would put the patient at increased risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with dose limiting toxicities evaluated according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Up to 9 weeks after the initial dose of combination therapy
  The proportion of subjects who experienced grade ≥3 toxicities will be estimated, along with 95% confidence intervals by each type of toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lim, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No